CLINICAL TRIAL: NCT02270476
Title: Longitudinal Observational Study on the Course of Cystic Fibrosis Lung Disease in Patients Following Newborn Screening
Acronym: TRACK-CF
Status: Recruiting | Type: Observational
Sponsor: Heidelberg University (Other)
Collaborators: German Center for Lung Research (Other)
Responsible Party: Principal Investigator, Mirjam Stahl, PI and Leader of Junior Research Group, Heidelberg University
Other Study IDs: UKH-TRACK-1
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Cystic Fibrosis Lung Disease
Keywords: Cystic Fibrosis; Infant; Toddler; Children; Newborn screening
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early diagnosed (ED): Children diagnosed with CF in the first 4 months of life.
- Late diagnosed (LD): Children diagnosed with CF after the first 4 months of life.

SUMMARY:
The purpose of this study is to further characterize early CF lung disease in newborns, infants and toddlers with cystic fibrosis (CF).

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most common lethal genetic multisystem disease in Germany. Although life expectancy increased over the last decades, most of the CF patients die in young adulthood due to chronic CF lung disease with respiratory failure. CF lung disease is caused by a disturbed transport of salt and water by airway epithelia and dehydration of airway surfaces as a result of the underlying genetic defect in the Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) gen. Up to now, no causal therapies for the majority of patients with CF are available. Little is known about onset and natural course as well as influencing factors of CF lung disease. Therefore, the first aim of this prospective, multicenter, uncontrolled, non-randomized, explorative longitudinal study is characterization of the onset and early course of CF lung disease. For this reason we will primarily include patients diagnosed by CF newborn screening (CF-NBS) or for any other reason in the first four months of life (early diagnosed, ED). In a second step we will compare data from these patients to those diagnosed clinically later in life (late diagnosed, LD). This will allow us to investigate the effect of early diagnosis and start of therapy. Starting at diagnosis, we will use data from annual routine check-ups (imaging like chest MRI, pulmonary function tests, microbiology from swabs and sputum, laboratory values, anthropometry) as well as data from a facultative, study-related bronchoscopy with lavage (microbiology, inflammation and immunology) for correlation with the course of CF lung disease (generation of hypotheses). Further study-related investigations are monthly telephone interviews on bronchopulmonary symptoms by a study nurse on the basis of a questionnaire and quarterly assessment of health-related quality of life on the basis of a validated questionnaire.

We expect to gain a deeper insight into onset and early course of CF lung disease from the results of this study. So far, there is no trial that investigated the different aspects of CF lung disease (function, morphology, infectiology, inflammation) complementary in a longitudinal setting. We assume that knowledge on the natural history of CF lung disease in the vulnerable phase of early childhood has a great impact on the future development of new therapies (from symptomatic to causal). This shall lead to a further improvement in life expectancy and quality of life of patients with CF.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed patients with Cystic Fibrosis (CF). Diagnosis of CF: at least one of the following three international accepted criteria is fulfilled: i) sweat chloride ≥ 60mEq/L and/or ii) 2 CF-causing mutations in the CFTR gene and/or iii) changes typical for CF in the transepithelial potential difference in nasal or rectal epithelium.
2. Age and mode of diagnosis:

   * Early diagnosed (ED): Initial diagnosis following CF-NBS or for other reasons in the first 4 months of life (in preterms corrected age of 4 months) after January 1st, 2006. Other reasons could be prenatal diagnostics, meconium ileus or positive family history.
   * Late diagnosed (LD): Diagnosed after the fourth month of life due to clinical symptoms; initial diagnosis after January 1st, 2006.

Exclusion Criteria:

All patients are excluded who themselves or whose parents do not want to participate or that withdraw from the study; or those in whom the diagnosis of CF is unsure.

Further exclusion criteria are:

1. Preterms <30th week of gestation
2. Longer period of mechanical ventilation in first 3 months of life
3. A significant medical disease or condition other than CF likely to interfere with the child's ability to complete the entire protocol
4. Previous major surgery except for meconium ileus or atresia of the intestine
5. Other major organ dysfunction, excluding pancreatic or hepatic dysfunction or another condition due to CF
6. Physical findings that would compromise the safety of the subject or the quality of the study data as determined by investigator
7. Chronic lung disease other than CF (e.g. bronchopulmonary dysplasia)
8. History of adverse reaction to medication for sedation or known claustrophobia

Criteria, which lead to a displacement of the procedures in sedation until the child has recovered: - Clinically significant upper airway obstruction as determined by investigator (e.g.

severe laryngomalacia, markedly enlarged tonsils, significant snoring, diagnosed obstructive sleep apnoea)

- Severe gastroesophageal reflux, defined as persistent frequent emesis despite anti-reflux therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CF diagnosed in the first 4 months of life (corrected age of 4 months in preterms) not before January 1st, 2006 build up the early diagnosed (ED) group. Early identification can be achieved by newborn screening, clinical diagnosis (e.g. patients with meconium ileus), due to positive family history or prenatal diagnosis. Patients with CF diagnosed after the first 4 months of life and after January 1st, 2006, are included as a comparison group with clinically diagnosed patients (late diagnosed, LD). Both groups (ED and LD) are investigated after the same investigational plan with all investigations that are part of the annual check-up and additional, study-related monthly telephone interviews on bronchopulmonary symptoms, quarterly assessment of QoL and voluntarily yearly bronchoscopy with broncho-alveolar lavage.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-12; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Proportion with morphological and/or perfusion changes due to CF lung disease after chest MRI score in both groups | At age of 1, 2, 3, ...., 10 years of age
Proportion of patients with impairments in pulmonary function tests (e.g. multiple breath washout (MBW)) in both groups | At age of 1, 2, 3, ...., 10 years of age

SECONDARY OUTCOMES:
Rate of protocol-defined pulmonary exacerbations in both groups (ED vs. LD) that are necessitating an antibiotic therapy orally, intravenously or per inhalation | At age of 1, 2, 3, ...., 10 years of age
Spontaneous development of infection or spectrum of pathogens, respectively, in throat and nose swabs as well as other airway secretions from routine diagnostics and if applicable bronchoalveolar lavage fluid (BALF) | At age of 1, 2, 3, ...., 10 years of age
From the patients in whom PsA or other CF pathogens could not be isolated at the beginning of their participation, comparison of the portion of patients with a positive culture during participation in both groups (ED and LD) | At age of 1, 2, 3, ...., 10 years of age
Time to first detection of a CF pathogen in both groups | At age of 1, 2, 3, ...., 10 years of age
Time to first pulmonary exacerbation in both groups | At age of 1, 2, 3, ...., 10 years of age
Portion of patients with increased biochemical inflammatory markers in both groups and magnitude of elevation | At age of 1, 2, 3, ...., 10 years of age
Frequency of symptoms from monthly telephone interviews in both groups | At age of 1, 2, 3, ...., 10 years of age
Health-related quality of life in both groups quarterly via Cystic Fibrosis Questionnaire (CFQ) | At age of 1, 2, 3, ...., 10 years of age
Development of body weight, body height, ideal weight-for-height (IWFH), Body-Mass-Index (BMI), respiratory rate and oxygen saturation at room air in both groups | At age of 1, 2, 3, ...., 10 years of age
Proportion with morphological changes due to CF lung disease after modified Chrispin-Norman Score for assessment of chest X-ray in both groups | At age of 1, 2, 3, ...., 10 years of age
Magnitude and severity of alterations typical for CF by assessment with chest MRI and X-ray score in both groups | At age of 1, 2, 3, ...., 10 years of age
Magnitude of impairment of pulmonary function test in both groups | At age of 1, 2, 3, ...., 10 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Marcus A Mall, MD, Principal Investigator — University Hospital Heidelberg
Locations (4):
- Germany (4):
  - University Children's Hospital Heidelberg, Cystic Fibrosis Centre, Heidelberg, Baden-Wurttemberg
  - University Hospital Gießen and Marburg GmbH, Giessen, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - University Children's Hospital Schleswig-Holstein, Lübeck, Schleswig-Holstein

REFERENCES:
- [Derived] Wielputz MO, Stahl M, Triphan SMF, Wucherpfennig L, Leutz-Schmidt P, Gestewitz S, Steinke E, Graeber SY, Kauczor HU, Eichinger M, Puderbach MU, Alrajab A, Schenk JP, Sommerburg O, Mall MA. Longitudinal Magnetic Resonance Imaging of Changes in Lung Morphology and Perfusion in Children with Cystic Fibrosis from Infancy through Adolescence. Ann Am Thorac Soc. 2025 Jan;22(1):93-103. doi: 10.1513/AnnalsATS.202404-396OC. PMID 39255452
- [Derived] Steinke E, Sommerburg O, Graeber SY, Joachim C, Labitzke C, Nissen G, Ricklefs I, Rudolf I, Kopp MV, Dittrich AM, Mall MA, Stahl M. TRACK-CF prospective cohort study: Understanding early cystic fibrosis lung disease. Front Med (Lausanne). 2023 Jan 6;9:1034290. doi: 10.3389/fmed.2022.1034290. eCollection 2022. PMID 36687447
- [Derived] Wucherpfennig L, Wuennemann F, Eichinger M, Schmitt N, Seitz A, Baumann I, Stahl M, Graeber SY, Chung J, Schenk JP, Alrajab A, Kauczor HU, Mall MA, Sommerburg O, Wielputz MO. Longitudinal Magnetic Resonance Imaging Detects Onset and Progression of Chronic Rhinosinusitis from Infancy to School Age in Cystic Fibrosis. Ann Am Thorac Soc. 2023 May;20(5):687-697. doi: 10.1513/AnnalsATS.202209-763OC. PMID 36548543
- [Derived] Stahl M, Steinke E, Graeber SY, Joachim C, Seitz C, Kauczor HU, Eichinger M, Hammerling S, Sommerburg O, Wielputz MO, Mall MA. Magnetic Resonance Imaging Detects Progression of Lung Disease and Impact of Newborn Screening in Preschool Children with Cystic Fibrosis. Am J Respir Crit Care Med. 2021 Oct 15;204(8):943-953. doi: 10.1164/rccm.202102-0278OC. PMID 34283704
- [Derived] Stahl M, Wielputz MO, Graeber SY, Joachim C, Sommerburg O, Kauczor HU, Puderbach M, Eichinger M, Mall MA. Comparison of Lung Clearance Index and Magnetic Resonance Imaging for Assessment of Lung Disease in Children with Cystic Fibrosis. Am J Respir Crit Care Med. 2017 Feb 1;195(3):349-359. doi: 10.1164/rccm.201604-0893OC. PMID 27575911